CLINICAL TRIAL: NCT00225212
Title: Clinical Trial Of C2B8 Monoclonal Antibody Following High Dose Therapy And Autografting In B-Cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab After Autologous Stem Cell Transplant for Relapsed B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: protocol97; 73750 (Other: Stanford IRB, old system)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Non-Hodgkin's Lymphoma; Diffuse Large Cell Lymphoma; Mantle Cell Lymphoma; Transformed Lymphoma; Other Subtypes of B-cell Lymphoma; Lymphoma
Keywords: non-Hodgkin's lymphoma; diffuse large cell lymphoma; mantle cell lymphoma; transformed lymphoma; other subtypes of B cell lymphoma; recurrent lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab after ASCT (Experimental): Rituximab 375 mg/m2 starting 6 weeks after ASCT transplant, and for the 5th and subsequent subjects, a second course at the same dose 6 months after ASCT.
  Interventions: Drug: Rituximab 375 mg/m2

INTERVENTIONS:
Drug: Rituximab 375 mg/m2
  Other Names: Rituxan; MabThera; Zytux; IDEC-C2B8; chimeric anti-CD20

SUMMARY:
Conventional therapy is effective for diffuse aggressive lymphomas and low grade lymphomas, but is limited by relapse occurs in 40 to 50% of subjects.

This study assesses autologous stem cell transplant (ASCT) supplemented with high-dose therapy increases the event-free survival in diffuse aggressive lymphomas and low grade lymphomas, as an alternative to the limitations of conventional therapy.

Preliminary studies with rituximab in low grade lymphomas indicate a response rate of about 50% with very little toxicity. Rituximab is hypothesized to be a candidate for post-transplant therapy because the majority of malignant lymphomas express the CD20 antigen; rituximab has impressive independent anti-tumor activity; and the antibody has little toxicity outside of the acute administration.

DETAILED DESCRIPTION:
The first 4 subjects received rituximab weekly for 4 weeks at the standard dose of 375 mg/m2, starting 6 weeks after ASCT transplant.

After an observation period to assess acute and late toxicity for the first 4 subjects, subsequent subjects received induction as above followed by an additional 4 week course at 6-months post-ASCT.

ELIGIBILITY:
Inclusion Criteria:

* B-cell, CD20+ NHL
* Evidence of engraftment post-autologous peripheral blood stem cell transplant (PBSC-T), aka autologous stem cell transplant (ASCT)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Creatinine < 2 mg/dL
* Bilirubin < 2.0 mg/dL
* Liver function tests (LFTs) < 5 x upper limit of normal (ULN)

Exclusion Criteria:

* Graft source from bone marrow
* Non-responders [progressive disease (PD) or stable disease (SD)] to prior anti-CD20 therapy
* PD after ASCT
* Post-ASCT radiotherapy
* Concomitant treatment with radiotherapy, chemotherapy or immunotherapy including rituximab
* Evidence of active pneumonitis
* Evidence of active infection
* Concurrent prednisone or other systemic steroid medication
* Nitrosourea therapy within 6 weeks of the first treatment with rituximab
* Presence of anti-murine antibody (HAMA) reactivity

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1997-11; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J Horning, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Result] Horwitz SM, Negrin RS, Blume KG, Breslin S, Stuart MJ, Stockerl-Goldstein KE, Johnston LJ, Wong RM, Shizuru JA, Horning SJ. Rituximab as adjuvant to high-dose therapy and autologous hematopoietic cell transplantation for aggressive non-Hodgkin lymphoma. Blood. 2004 Feb 1;103(3):777-83. doi: 10.1182/blood-2003-04-1257. Epub 2003 Aug 7. PMID 12907446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab After ASCT
Started | 35
Completed | 29
Not Completed | 6
Not completed — Disease progression | 2
Not completed — Death | 1
Not completed — Adverse Event | 2
Not completed — Intercurrent illness | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab After ASCT
Number analyzed (Participants) | 35
Age, Customized [Median (Full Range); unit: years] — B-cell lymphoma patients aged 16 and older
  years
    aged 16 and older | 51 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 23
Lymphoma sub-types [Number; unit: participants]
  Diffuse large B-cell lymphoma (DLCL) | 25
  Mantle cell lymphoma (MCL) | 3
  Transformed lymphoma | 3
  Other B-cell lymphoma | 4

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: "Events" for EFS were defined as the earlier of post-ASCT relapse or death.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of not experiencing EFS event
Arm/Group | Rituximab After ASCT
Number analyzed (Participants) | 35
percentage of not experiencing EFS event | 83 [70 to 95]

2. Secondary Outcome: Overall Survival (OS)
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects remaining alive
Arm/Group | Rituximab After ASCT
Number analyzed (Participants) | 35
percentage of subjects remaining alive | 88 [78 to 99]

ADVERSE EVENTS:
Arm/Group | Rituximab After ASCT
Serious Adverse Events (participants affected / at risk) | 33/35
Other Adverse Events (participants affected / at risk) | 9/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab After ASCT (N=35)
Blood and lymphatic system disorders - Other, neutropenia (Blood and lymphatic system disorders) | 19 (45)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonitis, BCNU-related (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Death NOS, pneumonitis (General disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab After ASCT (N=35)
Blood and lymphatic system disorders - Other, neutropenia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic system disorders - Other, Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes